CLINICAL TRIAL: NCT00503477
Title: A Phase I Open Label Dose Escalation Study for the Safety and Tolerability of AZD2171 Following Single and Multiple Oral Doses in Patients in Japan With Advanced Solid Malignancies
Brief Title: A Phase I Open Label Dose Escalation Study for the Safety and Tolerability of AZD2171 in Solid Tumors in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jane Robertson, Medical Science Director,, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00023
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Advanced Solid Tumor
Keywords: Japan; Phase I; solid tumor; AZD2171
MeSH Terms: interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD2171 — oral tablet
  Other Names: cediranib; RECENTIN™

SUMMARY:
A Phase I open label dose escalation study to assess the safety and tolerability of AZD2171 following single and multiple oral doses in patients in Japan with advanced solid malignancies. In addition there will be an expanded cohort multi-centre study phase with NSCLC patient and CRC patients

ELIGIBILITY:
Inclusion Criteria:

* advanced solid tumors
* life expectancy is 12 weeks or longer

Exclusion Criteria:

* patient with uncontrolled brain metastases
* patient with inappropriate laboratory test values
* patient with poorly controlled hypertension

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Assessed at each visit for 4 weeks

SECONDARY OUTCOMES:
efficacy, PK | Assessed at each visit for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca; Tomohide Tamura, MD, Principal Investigator — National Cancer Centre Hospital, Tokyo
Locations (2):
- Japan (2):
  - Research Site, Shizuoka
  - Research Site, Tokyo